CLINICAL TRIAL: NCT06850116
Title: Analysis of Immediate Urinary Continence Predictors After Retzius-sparing Robot-assisted Radical Prostatectomy: A Single-center Retrospective Clinical Study
Brief Title: Analysis of Immediate Urinary Continence Predictors After RS-RARP
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MRCTA,ECFAH OfFMUI2025]002
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer (Post Prostatectomy); Urinary Continence; Retzius-sparing Robot-assisted Radical Prostatectomy
Keywords: Retzius-sparing robot-assisted radical prostatectomy; Prostate Cancer; urinary continence
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The Retzius-sparing robot-assisted radical prostatectomy group: In 2010, Italian urologist Dr Bocciardi carried out the first clinical practice of separation and resection of the prostate via the vesicorectal fossa, and this new surgical procedure was called Retzius-sparing Robotic Assisted Radical Prostatectomy (RS-RARP). In recent years, the posterior approach extrafascial technique of RS-RARP which has been used to widely resect the prostate and its surrounding fascia and neurovascular bundles, compared with RS-RARP, has been proposed to provide more complete resection of the tumour and reduce the rate of positive margins. The patients are included into the Retzius-sparing robot-assisted radical prostatectomy group group who undergo the posterior approach extrafascial technique of RS-RARP.
  Interventions: Procedure: Retzius-sparing robot-assisted radical prostatectomy

INTERVENTIONS:
Procedure: Retzius-sparing robot-assisted radical prostatectomy — Retzius-sparing robot-assisted radical prostatectomy

SUMMARY:
This study is a retrospective, single-center clinical trial. It aims to retrospectively analyze the immediate postoperative urinary continence recovery in prostate cancer patients who underwent Retzius-sparing robot-assisted radical prostatectomy in the investigators' center. Based on the general conditions of patients, relevant perioperative clinical indicators, and parameters related to the sphincter and prostate gland measured by MRI, it explores the influencing factors of immediate urinary continence recovery after Retzius-sparing robot-assisted radical prostatectomy in prostate cancer patients and constructs a relevant prediction model, thereby providing clinical guidance value for predicting immediate postoperative urinary continence recovery.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer diagnosed by prostate biopsy and underwent Retzius-sparing robot-assisted radical prostatectomy in the investigators' hospital.
* Received plain and contrast-enhanced pelvic or prostate MRI examinations before surgery.
* Eastern Cooperative Oncology Group (ECOG) performance status score between 0 and 1.
* Complete clinicopathological data.
* In good general condition, without infections, autoimmune diseases, hematological diseases or other malignant tumors.
* Complete postoperative follow-up data, with a postoperative follow-up time of no less than 6 months.

Exclusion Criteria:

* The patient has surgical contraindications.
* The patient has contraindications for MRI examination.
* Preoperative presence of congenital urinary system malformations, urinary incontinence or severe lower urinary tract symptoms, and with a history of urinary catheter or previous transurethral resection of the prostate (TURP) surgery.
* Having received neoadjuvant treatments that may affect the results of this study, such as radiotherapy or hormonal therapy.
* The patient has other concurrent malignant tumors.
* The patient has delayed extubation (> 14 days).
* The patient's clinical, imaging and pathological data are incomplete or the patient is lost to follow-up.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Prostate cancer patients underwent RS-RARP.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
rate of continence | rate of the preservation of urinary control function at 1 week after postoperative removal of the urinary catheter status
  Time Frame: 1 week after postoperative removal of the urinary catheter

CONTACTS AND LOCATIONS:
Locations (1):
- first hospital affiliated of Fujian medical university, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided